CLINICAL TRIAL: NCT05725993
Title: Longitudinal Assessment of Traumatic Microvascular Injury-2
Acronym: LATMI-2
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 852096
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI Patient
- Healthy Control

SUMMARY:
The goal of this observational study is to learn about changes in the brain of patients over the first 3 years following a traumatic brain injury (TBI). The main question it aims to answer are:

- How TBI effect the rate of brain tissue loss compare to healthy brain

Participants will give blood samples, complete MRI scans, and neuropsychological assessment measures.

Researchers will compare results between healthy control group and TBI group to determine changes in injured brains.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, inclusive
2. History of non-penetrating TBI of at least moderate severity (defined by evidence of trauma-related neuroimaging abnormality on cranial computerized tomography (CT) scan.
3. High-velocity, high-impact injury mechanism consistent with diffuse axonal injury (e.g., motor vehicle accident, fall from height, etc.)
4. Immediate loss of consciousness (cases with delayed loss of consciousness due to expanding lesions will be excluded)

Exclusion Criteria:

1. History of premorbid disabling neurological or psychiatric disease (such as epilepsy, brain tumors, meningitis, cerebral palsy, encephalitis, brain abscesses, vascular malformations, cerebrovascular disease, Alzheimer's disease, multiple sclerosis, HIV-encephalitis)
2. History of premorbid disability condition that would interfere with outcome assessments
3. Bilaterally absent pupillary Reponses
4. Penetrating TBI
5. Elevated intracranial pressure (≥ 17 mmHg) 6 Contradictions to contrast-enhanced MRI (e.g., ferromagnetic implants, pregnancy, allergy to gadolinium contrast, renal impairment [GFR < 60ml/g/m3], claustrophobia, hemodynamic instability)

7. Prisoners, patients in police custody 8. Objective lung disease (PaCO2 at rest > 50 mmHg or venous serum bicarbonate > 26 mEg/L) based on any labs available for review from patient's clinical care. Note that these will not be checked solely for study purposes 9.Requiring portable oxygen at enrollment 10. Chronic heart failure, severe pulmonary disease 11. Current substance abuse that precludes participation and follow-up in the study, as determined by the study investigators 12. If there is medical or other disability that precludes completion of the study procedures as determined by the study investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TBI subjects will be recruited directly from University of Pennsylvania Health System during their hospital stay. Healthy control subjects will be recruited via clinical practices, referring physicians, advertisements, Penn media services, social media avenues, iConnect, and community flyer.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Brain Atrophy | 3 years
  Rate of brain tissue volume loss quantified from serial brain MRI examinations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States